CLINICAL TRIAL: NCT03846349
Title: Non-invasive Reinforcement of the Upper Airway Dilator Muscles as an Alternative Approach to Treat Patients With Obstructive Sleep Apnea
Brief Title: Reinforcement of Upper Airway Muscles in Patients With OSAS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Haute Ecole de Santé Vaud (Other)
Responsible Party: Principal Investigator, Olivier Contal, Principal Investigator, Haute Ecole de Santé Vaud
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UAW strenghtening in OSAS
Record Dates: First submitted 2019-01-21; First posted 2019-02-19 (Actual); Last update posted 2019-10-28 (Actual); Status verified 2019-09

CONDITIONS: Obstructive Sleep Apnea Syndrome
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study Group (Experimental): Participants from the study group will follow an upper airway reinforcement regimen using the IOPI device over 6 weeks. The reinforcement protocol will be adapted each week to improve Percentage of initial strength Exercises will be adapted each week
  Interventions: Device: IOPI
- Control group (Sham Comparator): Participants from the control group will perform a sham reeducation protocol using an "EMT threshold" at minimal resistance. The expiratory pressure will remain unchanged over the weeks.
  Interventions: Device: EMT threshold

INTERVENTIONS:
Device: IOPI — IOPI is a portable device with a tongue bulb used to reinforce upper airway muscles.
  Arms: Study Group
Device: EMT threshold — EMT threshold is a small portable device producing a positive expiratory pressure when the patient is exhaling.
  Arms: Control group

SUMMARY:
This study will investigate the effectiveness of a simple and quick myofunctional reeducation protocol of the tongue in reducing the obstructive sleep apnea syndrome (OSAS) severity.

DETAILED DESCRIPTION:
This is a randomized controlled study. Participants with moderate OSAS severity will be either allocated to receive a myofunctional reeducation protocol (study group) or a sham protocol (control group). Apnea-hypopnea index (AHI) will be measured before and at the end (6 weeks) of the protocol. Participants from the study group will follow an upper airway reinforcement regimen using the IOPI (Iowa Oral Performance Instrument) device over 6 weeks while participants from the control group will perform a sham reeducation protocol using an "EMT threshold" at minimal resistance.

ELIGIBILITY:
Inclusion Criteria:

* Moderate obstructive sleep apnea syndrome (AHI between 15 and 30 events per hour)
* Poor adherence to continuous positive airway pressure (< 4h per night)

Exclusion Criteria:

* Craniofacial malformation
* Use of hypnotic medication
* Had stroke in the past
* Present a concurrent neuromuscular or severe obstructive nasal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-03-01 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in AHI (apnea-hypopnea index) on polygraphy | Baseline and 6 weeks
  Evolution of the number of apnea-hypopnea events (AHI) over 6 weeks. The AHI value at discharge will be compared with the baseline value.

SECONDARY OUTCOMES:
Change in tongue strength using the IOPI device | Baseline and 6 weeks
  Evolution of tongue strength over 6 weeks. Tongue strength will be measured by asking the participants to squeeze the tongue bulb of IOPI as much as possible over 3 seconds. Three trials are accepted and the best value will be recorded (Pmax). Pmax at discharge will be compared with Pmax at baseline.
Change in tongue endurance using the IOPI device | Baseline and 6 weeks
  Evolution of tongue endurance over 6 weeks. Tongue endurance will be measured by asking the participants to sustain a tongue pressure against the IOPI bulb at 50% of Pmax. Endurance will be assessed by measuring the holding duration of 50% of Pmax. Holding duration at discharge will be compared with the value at baseline.

CONTACTS AND LOCATIONS:
Locations (2):
- Switzerland (2):
  - Ligue Pulmonaire Genevoise, Geneva
  - Haute Ecole de Santé Vaud (HESAV), Lausanne